CLINICAL TRIAL: NCT06208722
Title: Testing a Mobile App to Improve Toothbrushing Skills and Habits in Teens With Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Donald Chi, Professor: School of Dentistry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00018248; UG3DE033184 (NIH)
Record Dates: First submitted 2023-12-22; First posted 2024-01-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Autism
Keywords: Toothbrushing app; Clinical trial; Habit formation; Evidence based
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomly selected in the experimental and the control arm. Participants in the experimental arm will use the experimental app while those in the control arm will use the control app. Participants will receive all surveys in the same format and frequency in both arms.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Investigator and Outcomes Assessor will be blinded to allocation. Both arms will be described as interventions (educational versus behavioral). At the end of the trial children will be able to access the app in the other arm free of charge. The Outcomes Assessor (Statistician) will be masked to group assignment and unblinded only after the final analyses are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Children in the experimental arm will receive the same health education module as in the control arm. They will also receive a brief tutorial on additional app components in the form of a digital social story, which is an effective way to convey information to children with autism. Participants will be completing 26-item Behavioral Survey at 2 weeks, 1 month, 2 month, and 3 month. Participants will be using the app during toothbrushing 2x a day for 3 months under direct supervision of the caregiver.
  Interventions: Behavioral: Testing a Mobile App to Improve Toothbrushing Skills and Habits in Teens With Autism
- Control (Other): The control arm will consist of a 20-second health education module delivered through the control app that consists of a digital selfie mirror and a timer that matches the length of brushing time in the experimental app. Participants will be completing all the survey activities similar to that of the participants in the experimental arm.
  Interventions: Behavioral: Testing a Mobile App to Improve Toothbrushing Skills and Habits in Teens With Autism

INTERVENTIONS:
Behavioral: Testing a Mobile App to Improve Toothbrushing Skills and Habits in Teens With Autism — Information provided in arm descriptions.

SUMMARY:
The goal of this proposed trial will modify an existing toothbrushing app for teens with autism and compare toothbrushing outcomes with a control app. We have 2 specific aims:

* During the 2-year UG3 phase, we will use the Discover, Design+Build, and Test Framework to modify our existing app and pilot the intervention.
* During the 4-year UH3 phase, we will recruit 270 pre-adolescents and teens with autism ages 10 to 17 years, randomize participants to one of two arms, and compare outcomes.

Participants will asked to use the app, complete surveys on REDCap, participate in feedback interviews and focus groups. Behavior change in the experimental group will be compared with that in the control group.

DETAILED DESCRIPTION:
Adolescents with autism are at increased risk for tooth decay in part because of poor diet and toothbrushing habits. Effective ways to reduce added sugar intake have yet to be tested, but technologies exist to help improve toothbrushing. Mobile health apps are a promising but underutilized way to improve and enforce toothbrushing habits. Many adolescents with autism are enamored with technology and own devices that support apps. We propose a Stage II efficacy trial in modifying a toothbrushing app and inform behavior change in the target population.

ELIGIBILITY:
Inclusion Criteria:

* Child participants will have Autism Spectrum Disorder that will be confirmed by: (1) chart review by clinical staff at the recruitment sites to determine if the child meets the DSM-5 criteria for autism spectrum disorder; OR (2) affirmative caregiver response (YES) to the question, "Has a healthcare provider ever diagnosed your child with autism?"
* Willingness to take a CARS-2 [Childhood Autism Rating Scale-2], which will be administered by trained staff
* Child brushes independently [The child needs to be able to hold the toothbrush and move it around their teeth, mostly unassisted]
* Child uses touch screen devices (e.g.,smartphones or tablet)
* Ages 10 to 17 years at enrollment
* Caregiver and child able to communicate in English
* Caregiver age ≥18 years and able to provide informed consent in English
* Child and caregiver live in the same home
* Child has ready access to a mobile device with a front-facing camera onto which apps can be downloaded (iPad or iPhone with iOS 16.0+; Android tablet or phone with Android 13.0+)
* Family has a Wi-Fi or cellular data plan to allow app data to be transmitted, with confirmation of via tools like the Ookla Speed Test to help problem solve and ensure that app data can be transmitted

Exclusion Criteria:

• Children with autism younger than age 10 years will be excluded

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Toothbrushing distribution | 3 months
  The primary outcome is toothbrushing distribution, defined as the mean proportion of total tooth surfaces in the mouth that are brushed during the last month of the 3-month trial.

SECONDARY OUTCOMES:
Toothbrushing duration | 3 months
  Toothbrushing duration (mean number of seconds brushed per toothbrushing episode during the last month of the 3-month trial) and frequency (number of days during the last month of the 3-month trial in which the app was used at least twice/day).

OTHER OUTCOMES:
Exploratory Outcome - long term behavior change | 9 months
  Long-term behavior change measured using the 4-item Behavioral Automaticity Index
Exploratory Outcome - oral health quality of life | 9 months
  Oral health quality of life measured using two items from the Child Oral Health Impact Profile-Reduced (COHIP-SF 19)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Chi, DDS, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States